CLINICAL TRIAL: NCT02607852
Title: System for Feedback of Patient Reported Outcomes in Children With Burns
Brief Title: Feedback System of PROMS in Children With Burns
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Stephanie Romo (Other)
Responsible Party: Sponsor-Investigator, Stephanie Romo, Clinical Research Technician, Shriners Hospitals for Children
Organization: Shriners Hospitals for Children (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: BOS1501; 20170611 (Other: Western Institutional Review Board)
Record Dates: First submitted 2015-08-17; First posted 2015-11-18 (Estimated); Last update posted 2017-06-22 (Actual); Status verified 2017-06

CONDITIONS: Burns
Keywords: Patient Reported Outcomes Measure; Burns
MeSH Terms: conditions — Burns

STUDY DESIGN:
Intervention Model Description: Arm A: Patients 5-18 years old Arm B: Patients 0-4 years old
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (Other): Patients between the ages of 5-18 years. They will complete the 5-18 version of the BOQ on iPads or through the HTTPS Tonic link.
  Interventions: Device: iPads
- Arm B (Other): Patients between the ages of 0-4 years. They will complete the 0-4 version of the BOQ and appropriate Pediatric Symptom Checklists (i.e. baby or preschool) on iPads or through the HTTPS Tonic link.
  Interventions: Device: iPads

INTERVENTIONS:
Device: iPads — The current study will help determine if using Burn Outcomes Questionnaire and 17- item Pediatric Symptom Checklist (PSC-17) feedback data, collected on iPads or online, over the course of patient treatment will be useful for the physicians and ultimately impact the recovery of the patient.

SUMMARY:
The primary objective of the overall study is to determine the feasibility and usefulness of a feedback system that delivers BOQ results to physicians in "real time" during outpatient encounters using iPads.

DETAILED DESCRIPTION:
The primary objective of this pilot study is to ascertain the feasibility and usefulness of a feedback system that provides clinicians with parent-proxy reported outcomes measure data during routine outpatient encounters for burn treatment.

The secondary objective of this first phase of the study is to determine clinicians' and parents perception of the experience of completing the BOQ+P and/or the usefulness of the information that was provided to the clinician and parent/guardians(s). For this reason we will collect a brief debriefing questionnaire from physicians and another from parents.

ELIGIBILITY:
Inclusion Criteria:

* Children between the ages of 0 and 18 years of age, receiving outpatient burn care at Shriners Hospitals for Children - Boston with total body surface area burn of ≥ 5% and/or a burn injury to face, hands, feet or genitalia. English or Spanish speaking and literate

Exclusion Criteria:

* Clinician overriding a patient to serve on the study because of medical/psychiatric problems that might in the opinion of the clinician overwhelm the goals/purposes of the study.

Max Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 35 (Actual)
Dates: Start 2015-04-08 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2017-12-31 (Estimated)

PRIMARY OUTCOMES:
Responses to Clinician Debriefing Questionnaires | Participants will participate for the duration of one outpatient visit, an expected average of 3 hours.
  After viewing the BOQ feedback and seeing the patient, the clinicians will rate whether or not they found the BOQ+P data useful. The measure includes 5 Likert-Scale questions and 1 open-ended question that asks for their feedback about the system.

CONTACTS AND LOCATIONS:
Overall Officials: Robert L Sheridan, MD, Principal Investigator — Shriners Hospitals for Children
Locations (1):
- Shriners Hospitals for Children- Boston, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No